CLINICAL TRIAL: NCT02899299
Title: A Phase III, Randomized, Open Label Trial of Nivolumab in Combination With Ipilimumab Versus Pemetrexed With Cisplatin or Carboplatin as First Line Therapy in Unresectable Pleural Mesothelioma
Brief Title: Study of Nivolumab Combined With Ipilimumab Versus Pemetrexed and Cisplatin or Carboplatin as First Line Therapy in Unresectable Pleural Mesothelioma Patients
Acronym: CheckMate743
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-743; 2016-001859-43 (EudraCT Number)
Expanded Access: NCT02475382 (No longer available)
Record Dates: First submitted 2016-08-31; First posted 2016-09-14 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Nivolumab; Ipilimumab; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nivolumab and Ipilimumab (Experimental): Specified dose on specified days
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Pemetrexed and Cisplatin (or Carboplatin) (Active Comparator): Specified dose on specified days
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558; Opdivo
  Arms: Nivolumab and Ipilimumab
Biological: Ipilimumab
  Other Names: BMS-734016; Yervoy
  Arms: Nivolumab and Ipilimumab
Drug: Pemetrexed
  Arms: Pemetrexed and Cisplatin (or Carboplatin)
Drug: Cisplatin
  Arms: Pemetrexed and Cisplatin (or Carboplatin)
Drug: Carboplatin
  Arms: Pemetrexed and Cisplatin (or Carboplatin)

SUMMARY:
The purpose of this study is to test the effectiveness and tolerability of the combination of Nivolumab and Ipilimumab compared to Pemetrexed and Cisplatin or Carboplatin in patients with unresectable pleural mesothelioma.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Males and Females at least 18 years of age
* Histologically confirmed pleural malignant mesothelioma not eligible for curative surgery
* ECOG Performance status of 0 or 1
* Available tumor sample for testing
* Acceptable blood work

Exclusion Criteria:

* Primitive peritoneal, pericardial and tunica vaginalis testis mesotheliomas
* Prior chemotherapy for pleural mesothelioma
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2 oranti-CTLA-4 antibody
* History of other malignancy unless the subject has been disease-free for at least 3 years
* Active, untreated central nervous system (CNS) metastasis

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2023-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (109):
- United States (14):
  - Ucsf, San Francisco, California
  - Local Institution - 0014, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center & Research Inst, Inc, Tampa, Florida
  - Local Institution - 0002, Chicago, Illinois
  - Univ Of Maryland Greenbaum Cancer Center, Baltimore, Maryland
  - Local Institution - 0013, Detroit, Michigan
  - Cancer & Hematology Centers Of Western Michigan, Grand Rapids, Michigan
  - Local Institution - 0004, Rochester, Minnesota
  - Memorial Sloan Kettering Nassau, New York, New York
  - Local Institution - 0007, Cleveland, Ohio
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Local Institution - 0005, Houston, Texas
  - West Virginia University, Morgantown, West Virginia
- Australia (5):
  - Local Institution - 0032, Sydney, New South Wales
  - Local Institution - 0031, Birtinya, Queensland
  - Local Institution - 0033, Clayton, Victoria
  - Local Institution - 0030, Malvern, Victoria
  - Local Institution - 0034, Nedlands, Western Australia
- Belgium (4):
  - Local Institution - 0089, Brussels
  - Local Institution - 0086, Edegem
  - Local Institution - 0087, Liège
  - Local Institution - 0088, Sint-Niklaas
- Brazil (2):
  - Local Institution, Barretos, São Paulo
  - Local Institution - 0064, São Paulo
- Local Institution - 0018, Santiago, Santiago Metropolitan, Chile
- China (5):
  - Local Institution - 0133, Harbin, Heilongjiang
  - Local Institution, Changchun, Jilin
  - Local Institution, Shenyang, Liaoning
  - Local Institution - 0124, Kunming
  - Local Institution - 0120, Shanghai
- Colombia (2):
  - Local Institution - 0039, Bogotá
  - Local Institution - 0040, Bogotá
- France (10):
  - Local Institution - 0057, Caen
  - Local Institution - 0073, Créteil
  - Local Institution - 0074, La Tronche
  - Local Institution - 0067, Lille
  - Local Institution - 0069, Marseille
  - Local Institution - 0056, Paris
  - Local Institution - 0080, Saint-Herblain
  - Local Institution - 0093, Strasbourg
  - Local Institution - 0058, Toulon
  - Local Institution - 0068, Toulouse
- Germany (10):
  - Local Institution - 0026, Cologne
  - Local Institution - 0054, Coswig
  - Local Institution - 0038, Essen
  - Local Institution - 0023, Göttingen
  - Local Institution - 0024, Großhansdorf
  - Local Institution - 0027, Hamburg
  - Local Institution - 0037, Heidelberg
  - Local Institution - 0021, Homburg An D. Saar
  - Local Institution - 0022, Immenhausen
  - Local Institution - 0019, Moers
- Greece (2):
  - Local Institution - 0017, Athens
  - Local Institution - 0016, Thessaloniki
- Italy (8):
  - Local Institution - 0042, Ravenna, Emilia-Romagna
  - Local Institution - 0047, Aviano
  - Local Institution - 0044, Bari
  - Local Institution - 0046, Catania
  - Local Institution - 0045, Genova
  - Local Institution - 0043, Napoli
  - Local Institution - 0048, Rozzano
  - Local Institution - 0041, Siena
- Japan (15):
  - Local Institution - 0105, Nagoya, Aichi-ken
  - Local Institution - 0097, Chiba, Chiba
  - Local Institution - 0108, Fukuyama-shi, Hiroshima
  - Local Institution - 0114, Hiroshima, Hiroshima
  - Local Institution - 0101, Sapporo, Hokkaido
  - Local Institution - 0106, Amagasaki-shi, Hyōgo
  - Local Institution - 0098, Nishinomiya-shi, Hyōgo
  - Local Institution - 0095, Yokohama, Kanagawa
  - Local Institution - 0104, Natori-shi, Miyagi
  - Local Institution - 0107, Niigata, Niigata
  - Local Institution - 0100, Okayama, Okayama-ken
  - Local Institution - 0096, Kitaadachi-gun, Saitama
  - Local Institution - 0094, Chuo-ku, Tokyo
  - Local Institution - 0099, Ube-shi, Yamaguchi
  - Local Institution - 0113, Sayama
- Mexico (5):
  - Local Institution - 0051, Guadalajara, Jalisco
  - Local Institution - 0079, Df, Mexico City
  - Local Institution - 0053, Mexico City, Mexico City
  - Local Institution - 0050, Mexico City, Mexico City
  - Local Institution - 0118, Chihuahua City
- Netherlands (2):
  - Local Institution - 0092, Amsterdam
  - Local Institution - 0091, Rotterdam
- Poland (3):
  - Local Institution - 0078, Bytom
  - Local Institution - 0076, Krakow
  - Local Institution - 0077, Warsaw
- Romania (4):
  - Local Institution - 0115, Bucharest
  - Local Institution - 0109, Bucharest
  - Local Institution - 0102, Craiova
  - Local Institution - 0055, Romania
- Russia (3):
  - Local Institution - 0150, Moscow
  - Local Institution - 0071, Moscow
  - Local Institution - 0072, Saint Petersburg
- South Africa (2):
  - Local Institution - 0060, Pretoria, Gauteng
  - Local Institution - 0059, Cape Town, Western Cape
- Switzerland (3):
  - Local Institution - 0049, Bern
  - Local Institution - 0036, Lausanne
  - Local Institution - 0029, Zurich
- Turkey (Türkiye) (3):
  - Local Institution - 0111, Diyarbakır
  - Local Institution - 0112, Istanbul
  - Local Institution - 0110, Seyhan
- United Kingdom (6):
  - Local Institution - 0085, Truro, Cornwall
  - Local Institution - 0084, Edinburgh, Midlothian
  - Local Institution - 0081, Leicester
  - Local Institution - 0083, London
  - Local Institution - 0116, Manchester
  - Local Institution - 0090, Southampton

REFERENCES:
- [Derived] Scherpereel A, Antonia S, Bautista Y, Grossi F, Kowalski D, Zalcman G, Nowak AK, Fujimoto N, Peters S, Tsao AS, Mansfield AS, Popat S, Sun X, Lawrance R, Zhang X, Daumont MJ, Bennett B, McKenna M, Baas P. First-line nivolumab plus ipilimumab versus chemotherapy for the treatment of unresectable malignant pleural mesothelioma: patient-reported outcomes in CheckMate 743. Lung Cancer. 2022 May;167:8-16. doi: 10.1016/j.lungcan.2022.03.012. Epub 2022 Mar 21. PMID 35367910
- [Derived] Peters S, Scherpereel A, Cornelissen R, Oulkhouir Y, Greillier L, Kaplan MA, Talbot T, Monnet I, Hiret S, Baas P, Nowak AK, Fujimoto N, Tsao AS, Mansfield AS, Popat S, Zhang X, Hu N, Balli D, Spires T, Zalcman G. First-line nivolumab plus ipilimumab versus chemotherapy in patients with unresectable malignant pleural mesothelioma: 3-year outcomes from CheckMate 743. Ann Oncol. 2022 May;33(5):488-499. doi: 10.1016/j.annonc.2022.01.074. Epub 2022 Feb 3. PMID 35124183
- [Derived] Baas P, Scherpereel A, Nowak AK, Fujimoto N, Peters S, Tsao AS, Mansfield AS, Popat S, Jahan T, Antonia S, Oulkhouir Y, Bautista Y, Cornelissen R, Greillier L, Grossi F, Kowalski D, Rodriguez-Cid J, Aanur P, Oukessou A, Baudelet C, Zalcman G. First-line nivolumab plus ipilimumab in unresectable malignant pleural mesothelioma (CheckMate 743): a multicentre, randomised, open-label, phase 3 trial. Lancet. 2021 Jan 30;397(10272):375-386. doi: 10.1016/S0140-6736(20)32714-8. Epub 2021 Jan 21. PMID 33485464
- [Derived] Wright K. FDA Approves Nivolumab Plus Ipilimumab for Previously Untreated Unresectable Malignant Pleural Mesothelioma. Oncology (Williston Park). 2020 Nov 12;34(11):502-503. doi: 10.46883/ONC.2020.3411.0502. PMID 33206991
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT02899299.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A: Nivolumab 3 mg/kg IV Q2W + Ipilimumab 1 mg/kg IV Q6W
- Treatment B: Pemetrexed 500 mg/m^2 + Cisplatin 75 mg/m^2 or Carboplatin 5 AUC up to 6 cycles
Period: Pre-treatment
Arm/Group | Treatment A | Treatment B
Started (Started = Randomized) | 303 | 302
Completed (Completed = Entering treatment) | 300 | 284
Not Completed | 3 | 18
Not completed — Participant request to discontinue study treatment | 0 | 3
Not completed — Participant withdrew consent | 1 | 11
Not completed — Participant no longer meets study criteria | 2 | 3
Not completed — Not reported | 0 | 1
Period: Treatment
Arm/Group | Treatment A | Treatment B
Started (Started = Entering treatment) | 300 | 284
Completed (Completed) | 0 | 189
Not Completed | 300 | 95
Not completed — Disease Progression | 182 | 43
Not completed — Study Drug Toxicity | 60 | 24
Not completed — Adverse Event unrelated to Study Drug | 11 | 9
Not completed — Participant request to discontinue Study treatment | 4 | 10
Not completed — Participant withdrew consent | 6 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Maximum Clinical Benefit | 11 | 2
Not completed — Poor/Non-compliance | 1 | 0
Not completed — Participant no longer meets Study criteria | 4 | 0
Not completed — Administrative reason by Sponsor | 2 | 0
Not completed — Other reasons | 12 | 2
Not completed — Not reported | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Total
Number analyzed (Participants) | 303 | 302 | 605
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.7 (8.5) | 67.8 (9.7) | 68.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 69 | 138
  Male | 234 | 233 | 467
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 19 | 38
  Not Hispanic or Latino | 122 | 136 | 258
  Unknown or Not Reported | 162 | 147 | 309
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 26 | 39 | 65
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 266 | 250 | 516
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time from randomization to the date of death due to any cause. A participant who has not died was censored at last known date alive.
Time Frame: From randomization to the date of death (Up to 40 Months)
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 303 | 302
Months | 18.07 [16.82 to 21.45] | 14.09 [12.45 to 16.23]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority — Treatment A over Treatment B; p = 0.0020, Stratified Log Rank — Boundary for statistical significance was a p-value < 0.0345; This is 2 sided p-value from log-rank test stratified by histology and sex as entered in the IRT; Hazard Ratio (HR) = 0.74, 96.6% CI 2-sided [0.60 to 0.91] — Stratified Cox proportional hazard model

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate is defined as the percentage of randomized participants who achieve a best overall response of complete response (CR) or partial response (PR) per Blinded Independent Central Review (BICR) assessments. Per adapted m-RECIST for pleural mesothelioma, each single tumor measurement must be at least 10 mm in length to qualify as measureable disease and contribute to the sum that defines the pleural uni-variate measure. Per RECIST 1.1 for solid tumors, confirmation of response required:
  CR=Disappearance of all target lesions; PR=At least a 30% decrease in the sum of the Total Tumor Measurement; Progressive disease (PD)=At least a 20% increase in the sum of the Total Tumor Measurement.
Time Frame: From randomization date to the date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first (Up to 76 months)
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 303 | 302
Percentage of Participants | 39.3 [33.7 to 45.0] | 44.4 [38.7 to 50.2]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate is defined as the percentage of all randomized participants whose Best Overall Response was complete response (CR), partial response (PR), stable disease (SD) or Non-CR/Non-PD as assessed by Blinded Independent Central Review (BICR). Per adapted m-RECIST for pleural mesothelioma, each single tumor measurement must be at least 10 mm in length to qualify as measureable disease and contribute to the sum that defines the pleural uni-variate measure. Per RECIST 1.1 for solid tumors, confirmation of response required:
  CR=Disappearance of all target lesions; PR=At least a 30% decrease in the sum of the Total Tumor Measurement; Progressive disease (PD)=At least a 20% increase in the sum of the Total Tumor Measurement; SD=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Non-CR/Non-PD: Persistence of one or more non-target lesion(s).
Time Frame: From randomization date to the date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first (Up to 76 months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 303 | 302
Percentage of Participants | 76.6 [71.4 to 81.2] | 85.8 [81.3 to 89.5]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival is defined as the time between the date of randomization and the date of first documented tumor progression per Blinded Independent Central Review (BICR) assessments (using adapted m-RECIST and RECIST 1.1), or death due to any cause, whichever occurs first. Participants who received subsequent anticancer therapy prior to documented progression were censored at the date of the last evaluable tumor assessment conducted on or prior to the date of initiation of the subsequent anticancer therapy.
  Progressive disease (PD)=At least a 20% increase in the sum of the Total Tumor Measurement.
Time Frame: From randomization date to the date of first documented tumor progression or death due to any cause, whichever occurs first. (up to 76 months)
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 303 | 302
Months | 6.77 [5.59 to 7.36] | 7.23 [6.93 to 8.05]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority — Treatment A over Treatment B; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.77 to 1.13] — Stratified Cox proportional hazard model

5. Secondary Outcome: Overall Survival (OS) According to PD-L1 Expression Level
Description: PD-L1 Expression is defined as the percent of tumor cells membrane staining in a minimum of 100 evaluable tumor cells per validated Dako PD-L1 immunohistochemistry (IHC) assay. This is referred to as quantifiable PD-L1 expression and efficacy is determined by overall survival (OS) analysis. OS was defined as the time from randomization to the date of death due to any cause. A participant who has not died was censored at last known date alive.
Time Frame: From randomization date to the date of death (Up to 76 Months)
Population: All PD-L1 evaluable participants with baseline expression <1% or ≥1%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 289 | 297
Months
  <1% PD-L1: number analyzed (Participants) | 57 | 78
  <1% PD-L1 | 17.3 [10.1 to 23.9] | 16.6 [13.4 to 20.8]
  ≥1% PD-L1: number analyzed (Participants) | 232 | 219
  ≥1% PD-L1 | 18.0 [16.8 to 21.5] | 13.3 [11.6 to 15.4]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; <1% PD-L1; Test type: Superiority — Treatment A vs Treatment B; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.64 to 1.32]
Statistical Analysis 2: Comparison: Treatment A vs Treatment B; ≥1% PD-L1; Test type: Superiority — Treatment A vs Treatment B; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.59 to 0.88]

6. Secondary Outcome: Progression Free Survival (PFS) According to PD-L1 Expression Level
Description: PD-L1 Expression is defined as the percent of tumor cells membrane staining in a minimum of 100 evaluable tumor cells per validated Dako PD-L1 immunohistochemistry (IHC) assay. This is referred to as quantifiable PD-L1 expression and efficacy is determined by progression free survival (PFS) analysis. PFS is defined as the time between the date of randomization and the date of first documented tumor progression per Blinded Independent Central Review (BICR) assessments (using adapted m-RECIST and RECIST 1.1), or death due to any cause, whichever occurs first. Participants who received subsequent anticancer therapy prior to documented progression were censored at the date of the last evaluable tumor assessment conducted on or prior to the date of initiation of the subsequent anticancer therapy.
  Progressive disease (PD)=At least a 20% increase in the sum of the Total Tumor Measurement.
Time Frame: as for outcome 4
Population: All PD-L1 evaluable participants with baseline expression <1% or ≥1%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 289 | 297
Months
  <1% PD-L1: number analyzed (Participants) | 57 | 78
  <1% PD-L1 | 4.1 [2.7 to 5.6] | 8.3 [7.0 to 11.1]
  ≥1% PD-L1: number analyzed (Participants) | 232 | 219
  ≥1% PD-L1 | 7.0 [5.8 to 8.5] | 7.1 [6.2 to 7.6]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; < 1% PD-L1; Test type: Superiority — Treatment A vs Treatment B; Hazard Ratio (HR) = 1.79, 95% CI 2-sided [1.22 to 2.63]
Statistical Analysis 2: Comparison: Treatment A vs Treatment B; ≥1% PD-L1; Test type: Superiority — Treatment A vs Treatment B; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.61 to 0.96]

7. Secondary Outcome: Objective Response Rate (ORR) According to PD-L1 Expression Level
Description: PD-L1 Expression is defined as the percent of tumor cells membrane staining in a minimum of 100 evaluable tumor cells per validated Dako PD-L1 immunohistochemistry (IHC) assay. This is referred to as quantifiable PD-L1 expression and efficacy is determined by objective response rate (ORR) analysis. ORR is defined as the percentage of participants who achieve a best overall response of complete response (CR) or partial response (PR) per Blinded Independent Central Review (BICR) assessments. Per adapted m-RECIST for pleural mesothelioma, each single tumor measurement must be at least 10 mm in length to qualify as measureable disease and contribute to the sum that defines the pleural uni-variate measure.
  per RECIST 1.1 for solid tumors, confirmation of response required: CR=Disappearance of all target lesions; PR=At least a 30% decrease in the sum of the Total Tumor Measurement; Progressive disease (PD)=At least a 20% increase in the sum of the Total Tumor Measurement.
Time Frame: as for outcome 2
Population: All PD-L1 evaluable participants with baseline expression <1% or ≥1%
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 289 | 297
Percentage of Participants
  <1% PD-L1: number analyzed (Participants) | 57 | 78
  <1% PD-L1 | 21.1 [11.4 to 33.9] | 41.0 [30.0 to 52.7]
  ≥1% PD-L1: number analyzed (Participants) | 232 | 219
  ≥1% PD-L1 | 43.1 [36.6 to 49.7] | 45.7 [38.9 to 52.5]

8. Post Hoc Outcome: Extended Collection: Overall Survival (OS)
Description: as for outcome 1
Time Frame: From randomization date to the date of death (Up to 76 Months)
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 303 | 302
Months | 18.07 [16.82 to 20.99] | 14.09 [12.45 to 16.33]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority — Treatment A over Treatment B; p = 0.0008, Stratified Log Rank; This is 2 sided p-value from log-rank test stratified by histology and sex as entered in the IRT; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.62 to 0.88] — Stratified Cox proportional hazard model

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (up to approximately 76 months.) SAEs and Other AEs were assessed from first dose to 100 days post the last dose of study therapy (up to approximately 29 months).
Description: The number at Risk for All-Cause Mortality represents all randomized participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Groups:
- Nivolumab 3mg/kg Plus Ipilimumab 1mg/kg: Nivolumab 3 mg/kg IV Q2W + Ipilimumab 1 mg/kg IV Q6W
- Pemetrexed Plus Cisplatin or Carboplatin: Pemetrexed 500 mg/m^2 + Cisplatin 75 mg/m^2 or Carboplatin 5 AUC up to 6 cycles
Arm/Group | Nivolumab 3mg/kg Plus Ipilimumab 1mg/kg | Pemetrexed Plus Cisplatin or Carboplatin
All-Cause Mortality (participants affected / at risk) | 251/303 | 259/302
Serious Adverse Events (participants affected / at risk) | 188/300 | 106/284
Other Adverse Events (participants affected / at risk) | 277/300 | 264/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3mg/kg Plus Ipilimumab 1mg/kg (N=300) | Pemetrexed Plus Cisplatin or Carboplatin (N=284)
Anaemia (Blood and lymphatic system disorders) | 5 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 1
Myelosuppression (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Aortic valve disease (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Pleuropericarditis (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 4 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Opsoclonus myoclonus (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 9 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Overflow diarrhoea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Superior mesenteric artery dissection (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 1 | 2
Chest pain (General disorders) | 4 | 4
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 1
Hyperpyrexia (General disorders) | 2 | 0
Hyperthermia (General disorders) | 0 | 1
Illness (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 1
Mucosal inflammation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 4 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Performance status decreased (General disorders) | 0 | 1
Pyrexia (General disorders) | 16 | 4
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 5 | 0
Hepatitis (Hepatobiliary disorders) | 3 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 5 | 0
Contrast media allergy (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Infusion related hypersensitivity reaction (Immune system disorders) | 1 | 0
Abscess intestinal (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Candida sepsis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 1
Empyema (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Klebsiella urinary tract infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Otitis externa fungal (Infections and infestations) | 1 | 0
Pleural infection (Infections and infestations) | 2 | 1
Pleurisy bacterial (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 14 | 6
Pneumonia aspiration (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 51 | 42
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Limbic encephalitis (Nervous system disorders) | 2 | 0
Migraine (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0
Myasthenic syndrome (Nervous system disorders) | 1 | 0
Myelitis transverse (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 7 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 1
Renal haemorrhage (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
Giant cell arteritis (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3mg/kg Plus Ipilimumab 1mg/kg (N=300) | Pemetrexed Plus Cisplatin or Carboplatin (N=284)
Anaemia (Blood and lymphatic system disorders) | 41 | 118
Leukopenia (Blood and lymphatic system disorders) | 0 | 25
Neutropenia (Blood and lymphatic system disorders) | 5 | 79
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 32
Hypothyroidism (Endocrine disorders) | 37 | 3
Lacrimation increased (Eye disorders) | 1 | 19
Abdominal pain (Gastrointestinal disorders) | 30 | 13
Constipation (Gastrointestinal disorders) | 57 | 86
Diarrhoea (Gastrointestinal disorders) | 96 | 34
Nausea (Gastrointestinal disorders) | 76 | 124
Vomiting (Gastrointestinal disorders) | 47 | 55
Asthenia (General disorders) | 52 | 58
Chest pain (General disorders) | 22 | 21
Fatigue (General disorders) | 90 | 78
Malaise (General disorders) | 8 | 17
Non-cardiac chest pain (General disorders) | 39 | 16
Oedema peripheral (General disorders) | 47 | 19
Pain (General disorders) | 20 | 11
Pyrexia (General disorders) | 50 | 14
Nasopharyngitis (Infections and infestations) | 21 | 8
Infusion related reaction (Injury, poisoning and procedural complications) | 22 | 2
Alanine aminotransferase increased (Investigations) | 22 | 4
Amylase increased (Investigations) | 24 | 4
Blood alkaline phosphatase increased (Investigations) | 18 | 3
Blood creatinine increased (Investigations) | 26 | 19
Lipase increased (Investigations) | 27 | 4
Weight decreased (Investigations) | 17 | 24
Decreased appetite (Metabolism and nutrition disorders) | 72 | 75
Hypoalbuminaemia (Metabolism and nutrition disorders) | 19 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 19 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 9
Dizziness (Nervous system disorders) | 16 | 10
Dysgeusia (Nervous system disorders) | 15 | 22
Headache (Nervous system disorders) | 24 | 12
Neuropathy peripheral (Nervous system disorders) | 3 | 15
Insomnia (Psychiatric disorders) | 27 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 65 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 77 | 41
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 62 | 5
Rash (Skin and subcutaneous tissue disorders) | 60 | 21
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 | 5
Hypertension (Vascular disorders) | 16 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT02899299/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT02899299/SAP_001.pdf